CLINICAL TRIAL: NCT07299799
Title: Evidence-Based Nursing to Reduce Adverse Events Regarding Ventilator Associated Pneumonia, Pressure Injuries and Central Line Bloodstream Infection in Intensive Care Unit: A Quasi-experimental Study in Bangladesh
Brief Title: Evidence-Based Nursing to Reduce Adverse Events Regarding Ventilator Associated Pneumonia, Pressure Injuries and Central Line Bloodstream Infection in Intensive Care Unit in Bangladesh
Acronym: EBP in Nursing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Nahida Akhter, Principal Investigator, Ph.D Fellow, Graduate School of Biomedical and Health Sciences, Hiroshima University, Japan., Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BMRC/NREC/2025-2027/313; 65313072025 (Registry Identifier: BMRC (Bangladesh Medical Research Council)); 24K02733 (Registry Identifier: Japan Society for the Promotion of Science (JSPS))
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ventilator Acquired Pneumonia; Central Line Associated Blood Stream Infections (CLABSI); Pressure Ulcer (PU); Medical Device Related Pressure Ulcer (MDRPU)
Keywords: evidence based practice; Nurses competency; Ventilator Associated Pneumonia; Pressure Ulcer; Central Line Bloodstream Infection; Medical Device Related Pressure Ulcer
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pressure Ulcer | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Trial 1: A pre- and post- quasi-experimental study to evaluate the nurses competency (Skill, knowledge, practice and attitude).
  Trial 2: A pre- and post- quasi-experimental study to evaluate the outcomes of the patients in the ICU using study 1 Phase 1 data as historical data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Trial 1: All Nurses in GICU; Trial 2: All patients admitted in the general GICU (Experimental): Nurses: All nurses who work at GICU of DMCH Patients: all patients who will admit at the assigned GICU during the study period of DMCH
  Interventions: Behavioral: Education with EBP; Behavioral: This is a pre- and post- quasi-experimental study.

INTERVENTIONS:
Behavioral: Education with EBP — Trial 1: Nurse's EBP training ( VAP, PU, MDRPU, CLABSI management), online lecture, 2 hours lecture and 3 hours skill training for nurses training.
  Trail 1 we use advanced equipment necessary for EBP implementation for VAP, PU, MDRPU and CLABSI management, and EBP-trained nurses implementation for all this management.
Behavioral: This is a pre- and post- quasi-experimental study. — We will use advanced equipment and implement EBP (VAP, PU, MDRPU and CLABSI management) for patients by trained nurses and check the outcome of the patients. We will compare pre and post findings for this study.

SUMMARY:
Quality of care is crucial for preventing adverse events such as infection in the intensive care units (ICUs). The most common ICU-acquired infections include pneumonia such as Ventilator Associated Pneumonia (VAP), Pressure Ulcer (PU), Medical Device Related Pressure Ulcer (MDRPU), and Central Line-Associated Bloodstream Infection (CLABSI). VAP, PU, and MDRPU are significant indicators of the quality of care, while CLABSI is a critical marker of healthcare quality in ICUs, as it is largely preventable through strict adherence to infection control protocols.

VAP is a lung infection that occurs in patients receiving mechanical ventilation for more than 48 hours. A PU is defined as localized damage to the skin or underlying tissue caused solely by pressure, while MDRPUs may also result from friction or pressure from medical devices or other objects. CLABSI is a severe infection caused by improperly inserted or maintained central venous catheters, which underscores the need for stringent catheter management protocols.

DETAILED DESCRIPTION:
General Objective:

The objective of this study is to evaluate whether implementing EBP and changing nurses' competency (skill, knowledge, practice, and attitude) can reduce ICU adverse events such as VAP, PU, MDRPU, and CLABSI, and improve patient outcomes.

Specific Objectives:

1. To identify insights on perceptions, barriers, and facilitators related to EBP implementation in the ICU setting.
2. To evaluate the effect of EBP training on nurses' competency (skill, knowledge, practice, and attitude) regarding EBP for CLABSI, PU, and MDRPU in an ICU setting.
3. To evaluate the effects of EBP on ICU patient incidence rates of VAP, CLABSI, PU, and MDRPU.

Hypothesis:

H1- Hypothesize that training on EBP and its implementation in ICU settings will improve nurses' competency (Skill, knowledge, practice and attitude).

H2- Hypothesize that implementation of EBP by trained ICU nurses will reduce adverse events-such as VAP, pressure ulcers, medical device-related PU, and CLABSIs-and improve overall patient outcomes.

These research consist of two studies:

1. Evaluating the effect of EBP training on ICU nurses' competency (skill, knowledge, practice, and attitude) regarding EBP for CLABSI, PU, and MDRPU in an ICU setting.

   A pre- and post-quasi-experimental study will be conducted over a 16-month period, with a total data collection period of 6 months, to evaluate nurses' competency. The study consists of a recruitment period (1 month), nurses' baseline data collection (1 month), nurses' EBP training with midline data collection (2 months), and nurses' endline data collection during EBP implementation (2 months).

   Study nurses will receive EBP training and appropriate equipment for patient management. EBP education and training will be provided with necessary equipment, such as a closed suction catheter, an endotracheal tube, a suction device, and a mouth care brush. In this study, global standard equipment will be used to ensure patient safety.
2. Evaluating the effect of EBP implementation on ICU patient incidence rates of VAP, CLABSI, PU, and MDRPU.

A pre- and post-quasi-experimental design with a non-equivalent control group (Study 1, Phase 1 data used as historical data) will be applied by comparing the rate of adverse events such as VAP, CLABSI, PU, and MDRPU before and after the EBP intervention (2-month baseline data and 2-month intervention data will be collected).

ELIGIBILITY:
Trial 1 & 2-

Inclusion Criteria:

Nurse

* who is a registered nurse in Bangladesh.
* who agrees to participate in this study and the EBP training.
* who will stay at the ICU for 6 months. Patient
* Irrespective of age and sex, participants must be at least 18 years old
* Legal guardian of a patient consent to participation in the study

Exclusion Criteria:

Nurse

* Who will not directly involve patient care in ICU. Patient
* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The nurse's skill related to the PU, MDRPU and CLABSI total score measured by the researcher-developed checklist | 6 month data collection and total time frame of this study 16 months
  1. The nurse's skill and knowledge related to the PU, MDRPU and CLABSI checklist. Researcher developed checklist, 50 items with 0: not correct/did not do, 1: partially correct, 2: correct. Score range 0-114.
Incidence rates of PU, MDRPU and CLABSI. | 2 month for data collection and total time frame 16 months.
  The incidence rate of PU was calculated as the number of newly developed pressure ulcers after hospitalization per 1000 person-days at risk.
  The incidence rate of MDRPU was calculated as the number of newly developed MDRPU cases per 1000 patients assessed.
  The incidence rate of CLABSI was calculated as the number of CLABSI cases per 1000 central line-days.
  Data will be collected: Patients' demographic data (age, sex, occupation etc.) Medical past and current history (diagnosis, treatment, medication, hospitalization). Reasons and date to be admitted to ICU. Treatment in ICU. Daily laboratory data taken in ICU. Daily biological data including vital signs.
  Results of patients' stay during ICU. Diagnosis of PU, MDRPU and CLABSI included of this list.

SECONDARY OUTCOMES:
Nurses' knowledge, Attitude and Practice (KAP) related to the PU, MDRPU and CLABSI prevention measured by the researcher-developed scale based on Knowledge of EBP guidelines for the PU, MDRPU and CLABSI prevention scale | Total data collection time 6 months within 16 months
  Nurses attitude, practice and knowledge related PU, MDPU and CLABSI related prevention scale.
  The researcher makes an attitude, practice and knowledge related of EBP guideline for PU, MDPU and CLABSI question Total item 22 and validity was tested by ICU and PU specialized nurses in Japan.
  Knowledge was assessed using multiple-choice questions, with one correct answer among four options. Each correct response was awarded a score of 1, and incorrect or "don't know" responses were scored 0.
  Attitude and practice were measured using a Likert scale, with responses indicating the degree of agreement or frequency.
Rate (number of patients) of each stage of PU and MDRPU | Total 2 months
  After diagnosis of sore we measured stage of PU and MDRPU. Number of ICU patients developing PU and MDRPU categorized by stage (Stage I-IV). Unit of Measure: Number of patients per PU/MDRPU stage.
Micro-organism link to CLABSI | 2 months
  After diagnosis of CLABSI then identify what kind organism relate to CLABSI. Type and frequency of microorganisms identified in laboratory-confirmed CLABSI cases. Unit of Measure: Number of cases per microorganism.
Incidence and rate of VAP | 2 months
  Incidence rate of VAP per 1000 ventilator days. Unit of Measure: VAP cases per 1,000 ventilator days
Mortality and morbidity rate of adverse events | 2 months
  Mortality and morbidity rate of ICU patients All-cause mortality among ICU patients during the study period. Unit of Measure: Percentage (%)。Occurrence of ICU-related adverse events (VAP, CLABSI, PU, MDRPU). Unit of Measure: Number of patients with adverse events.
Average length of stay ICU patients | 2 months
  Average length of stay ICU patients. Mean length of stay in the intensive care unit for enrolled patients. Unit of Measure: Days (mean ± SD).
Survival rate of ICU | 2 months
  Average survival rate of ICU. Data will be collected: Length of stay and survival rate. Proportion of enrolled patients alive at ICU discharge. Unit of Measure: Percentage (%) of patients surviving to ICU discharge.

OTHER OUTCOMES:
APACHE II score | 2 months
  Will be collected from patient record file. Sum Acute Physiology Points + Age Points + Chronic Health Points = APACHE II total (range 0-71). APACHE II total score (integer). Optionally report distribution (mean ± SD) or stratify by score ranges.
SOFA score | 2 months
  Will be collected from patient record file. Sum Acute Physiology Points + Age Points + Chronic Health Points = APACHE II total (range 0-71). APACHE II total score (integer). Optionally report distribution (mean ± SD) or stratify by score ranges. Use worst values within first 24 h for baseline SOFA. For organ-dysfunction trajectory, compute daily SOFA scores。Sum component scores → SOFA total (0-24). SOFA total score (integer). Can also report number/proportion with increase ≥2 points.
GCS score | 2 months
  Total GCS = E + V + M (range 3-15). Record at ICU admission (worst value in first 24 h for scoring systems). Note if patient is sedated or intubated - document sedation/intubation; if intubated, record "V = T" and use local protocol for scoring (some protocols assign V=1 or use best pre-sedation score). Unit / reporting: GCS total (3-15). Report component scores if relevant.

CONTACTS AND LOCATIONS:
Locations (2):
- Dhaka Medical College Hospital, Dhaka, Dhaka Division, Bangladesh
- Hiroshima University, Hiroshima, Hiroshima City, Japan

IPD SHARING:
Plan to Share IPD: No
IPD will not be share due to personal confidentiality of the participants. When the data will be available and we will share the data according to the recommendations of the clinical trial registration and the requests of the journals.